CLINICAL TRIAL: NCT06798896
Title: RENAISSANCE 2: a Double-Blind, Randomized, Placebo-Controlled, Multicenter, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of SPN-817 in Adults with Focal Onset Seizures
Brief Title: RENAISSANCE 2: SPN-817 Phase 2, Double-Blind, Placebo-Controlled Study in Adults with Focal Onset Seizures
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 817P203
Record Dates: First submitted 2025-01-16; First posted 2025-01-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Focal Onset Seizures
Keywords: focal seizures; focal epilepsy; Phase 2; anti-seizure medication
MeSH Terms: conditions — Seizures; Epilepsies, Partial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPN-817 (Experimental): SPN-817, bid
  Interventions: Drug: SPN-817
- Placebo (Placebo Comparator): Placebo, bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPN-817 — SPN-817 starting at 0.25 mg bid up to 4.00 mg bid
  Arms: SPN-817
Drug: Placebo — Placebo, bid
  Arms: Placebo

SUMMARY:
This is a Phase 2 double-blind, randomized, placebo-controlled, multicenter, parallel-group study to evaluate the efficacy, safety, and tolerability of SPN-817 in adults with focal onset seizures.

DETAILED DESCRIPTION:
This is a Phase 2 double-blind, randomized, placebo-controlled, multicenter, parallel-group study to evaluate the efficacy, safety, and tolerability of SPN-817 administered as an adjunctive treatment in adults with focal onset seizures that have previously failed at least 2 anti-seizure medication (ASM) regimens. Participants will be taking 1 to 4 ASMs, with at least 4 seizures during the 6-week Screening Period. Following the Screening Period, eligible participants will be randomized 2:1 to SPN-817 (3.0-4.0 mg BID) or placebo and begin the Titration Period (8-10 weeks). In both treatment groups, open-label ondansetron (8 mg oral [PO]) will be taken prophylactically approximately 30 minutes before each SM dose (ie, BID) during the first 5 weeks of dose titration as an antiemetic; after the first 5 weeks, ondansetron may be taken as needed as either a preventative or therapeutic antiemetic. After the target dose of 3.0-4.0 mg BID is reached, participants will enter the Maintenance Period (14 weeks). Participants who complete the Maintenance Period will have the opportunity to enroll in a separate open-label study for continued treatment with SPN-817. Participants who do not enroll in the open-label study will undergo a Tapering Period (up to 4 weeks) and a follow-up safety phone call.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of treatment-resistant focal epilepsy as adjudicated by the Epilepsy Study Consortium, Inc (ESCI);
2. Failed to achieve sustained seizure freedom after ≥2 tolerated, appropriately chosen, and adequately dosed ASM drug schedules;
3. Able to keep accurate Seizure eDiaries (with the aid of a caregiver as needed);
4. Has a body mass index (BMI) between 18.0 and 40.0 kg/m2;
5. Treatment with a stable dose of 1 to 4 current ASMs for ≥28 days prior to screening. If following a diet plan along with the ASM, the participant should have been on a stable diet plan for at least 1 month prior to Visit 1. The diet plan should be maintained throughout the duration of the study;
6. At least 4 clinically observable focal onset seizures accepted by the ESCI prior to the first dose of SM (during the days of baseline Seizure eDiary data collection) and no more than a consecutive 21-day period that was seizure free. To be eligible for the study, participants must comply with the eDiary on at least 90% of the days of baseline data collection;

Exclusion Criteria:

1. Has taken huperzine A within the past 6 months;
2. Prior diagnosis of combined focal and generalized epilepsy syndrome as evidenced by severe developmental delay and multiple seizure types and confirmed by electroencephalography (EEG) (eg, Lennox-Gastaut syndrome). Participants should also be excluded in case of nondiagnostic information;
3. History of or current nonepileptic events that could be confused by the participant and/or study staff as epileptic seizures;
4. Only has seizures that are difficult to count; for example, seizures that are not clinically observable;
5. History of uncountable seizures, such as seizures that happen in a cluster that are too rapid to be counted individually;
6. History of status epilepticus within 6 months prior to screening;
7. Vagus nerve stimulation, deep brain stimulation, responsive neurostimulator system, or other neurostimulation for epilepsy device implanted or activated within 1 year prior to screening; or epilepsy surgery within 1 year prior to screening. Stimulation parameters for devices must have been stable for at least 3 months prior to Screening. Battery change for any epilepsy devices will be allowed; however, stimulation parameters must remain stable during the duration of the study;
8. Any suicidal behavior or suicidal ideation related to item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) based on the C-SSRS assessment in the 1 year before screening; a suicide attempt in the last 2 years before screening; or more than 1 lifetime suicide attempt;
9. Chronic concomitant therapy with non-ASMs that are cholinergic or anticholinergic.
10. History of >2 allergic reactions to an ASM or 1 serious hypersensitivity reaction to an ASM;
11. Any other reason which, in the opinion of the Investigator, would prevent the participant from taking part in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percent change (PCH) from baseline in focal onset seizure frequency per 28 days over the Maintenance Period | Baseline and Maintenance Period (Maintenance Week 1-14)
  Percent change in 28-day frequency of focal seizures during the 14 week Maintenance Period relative to baseline

SECONDARY OUTCOMES:
Proportion of subjects experiencing ≥50% reduction in focal seizure frequency per 28 days from baseline | Baseline and Maintenance Period (Maintenance Week 1-14)
  Greater than or equal to 50% reduction in 28-day frequency of focal seizures during the 14 week Maintenance Period relative to baseline.
PCH from baseline in focal onset seizure frequency per 28 days over the entire Treatment Period | Baseline through Titration Week 1 up to Week 10 and Maintenance Weeks 1-14
  Percent change in 28-day frequency of focal seizures during the entire Treatment Period (Titration Period + Maintenance Period) relative to baseline
Proportion of subjects experiencing ≥50% reduction in focal seizure frequency per 28 days from baseline | Baseline through Titration Week 1 up to Week 10 and Maintenance Weeks 1-14
  Greater than or equal to 50% reduction in 28-day frequency of focal seizures during the Treatment Period (Titration Period + Maintenance Period) relative to baseline.
Longest seizure-free interval over the entire Treatment Period | Baseline through Titration Week 1 up to Week 10 and Maintenance Weeks 1-14
  The longest intervals in days between two seizures during the entire Treatment Period.
Incidence of adverse events (AEs) | Baseline through Titration Week 1 up to Week 10, Maintenance Weeks 1-14, and Tapering Period up to Week 4
  The percent of subjects who took at least one dose of SPN-817 and reported at least one adverse event during SPN-817 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Himanshu Upadhyaya, MBBS, MS, MBA, Study Director — Supernus Pharmaceuticals, Inc.
Locations (1):
- Medsol Clinical Research Center, Port Charlotte, Florida, United States